CLINICAL TRIAL: NCT01155817
Title: A Phase 1 Study of Nilotinib in Steroid Dependent/Refractory Chronic Graft Versus Host Disease
Brief Title: Phase 1 Nilotinib in Steroid Dependent/Refractory Chronic Graft Versus Host Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, David Miklos, Assistant Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-18743; SU-06112010-6317 (Other: Stanford University); IRB-18743 (Other: Stanford IRB); BMT222 (Other: OnCore)
Record Dates: First submitted 2010-06-15; First posted 2010-07-02 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Bone Marrow Transplant Failure; Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Peripheral
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Peripheral | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — 200, 400, 800, oral
  Other Names: Tasigna; AMN107

SUMMARY:
PRIMARY OBJECTIVES:

Determine the safety and tolerability of nilotinib in steroid dependent / refractory cGVHD.

SECONDARY OBJECTIVES:

Determine the clinical efficacy of nilotinib in steroid dependent / refractory cGVHD.

ELIGIBILITY:
Inclusion Criteria:5.1.1 Steroid dependent/refractory cGVHD defined as:

1. Dependent disease - Persistent cGVHD manifestations requiring a glucocorticoid dose >= prednisone 0.25 mg/kg/day (0.5 mg/kg po qod) for at least 12 weeks.
2. Refractory disease - Progressive cGVHD manifestations despite treatment with a glucocorticoid dose >= prednisone 0.5 mg/kg/day (1 mg/kg po qod) for at least 4 weeks.

5.1.2 Any previous treatments for cGVHD (except nilotinib). Participants may have received nilotinib for other reasons besides cGVHD such as leukemia or solid tumor.

5.1.3 Participants must be receiving baseline systemic glucocorticoid therapy for cGVHD at study entry. The dose of steroids must be stable for 14 days prior to starting nilotinib.

5.1.4 At the time of trial enrollment, participants may be receiving one or two other immunosuppressive therapies in addition to glucocorticoids. Immunosuppressant doses must be stable for 14 days prior to starting nilotinib. Monoclonal T or B cell antibodies must be discontinued at least 28 days before starting nilotinib.

5.1.5 Chronic GVHD manifestations that can be followed on physical or laboratory exam. A list of potential manifestations is presented in Appendix D.

1. Skin changes
2. Oral mucosa changes
3. Hepatic dysfunction

5.1.6 >= 18 years old

5.1.7 Life expectancy >= 6 months.

5.1.8 Karnofsky performance status >= 60 (defined as being unable to work, able to live at home, and able to care for most personal needs but requiring occasional assistance from others).

5.1.9 Laboratory parameters:

1. Creatinine < 1.5 x ULN
2. ANC > 1.5 x 10^9/L
3. Platelets > 100 x 10^9/L
4. Total bilirubin < 1.5 x ULN
5. AST (SGOT) and ALT (SGPT) < 2.5 x ULN
6. Serum amylase and lipase <= 1.5 x ULN
7. Alkaline phosphatase <= 2.5 x ULN
8. Patients must have the following laboratory values within normal limits at the local institution lab or corrected to within normal limits with supplements prior to the first dose of study medication:

Potassium Magnesium Phosphorus Calcium

5.1.10 Oxygen saturation during exertion maintained at >= 88% on room air.

5.1.11 Ability to understand and willingness to sign a written informed consent form.

5.1.12 Females with reproductive potential must have a negative pregnancy test <= 7 days before starting nilotinib. Reproductive potential will be defined as having at least 1 menstrual period in the past 12 months. Male and female subjects with reproductive potential agree to the use of barrier contraception during their treatment and for up to 3 months after the last dose.

5.1.13 Careful rationalization of concomitant medications with the intent to discontinue or change to alternative medications when any concomitant medications are identified that have the potential to prolong the QTcB interval or are associated with an increased risk of torsades de pointes. (Appendix B)

5.1.14 . Careful rationalization of concomitant medications with the intent to discontinue or change to alternative medications if any concomitant medications are identified to be strong CYP3A4 inhibitors. (Appendix C)

5.1.15 Myeloablative or non-myeloablative allogeneic hematopoietic cell transplant.

Exclusion Criteria:5.2.1 Currently receiving or has received within 28 days of starting study drug nilotinib or any other tyrosine kinase inhibitor.

5.2.2 Received any anti-T or anti-B cell monoclonal antibody <= 28 days prior to the anticipated start of study drug.

5.2.3 Currently receiving > two immunosuppressants other than glucocorticoids.

5.2.4 Currently receiving a calcineurin inhibitor and sirolimus

5.2.5 Received any investigational agents <= 28 days before starting nilotinib.

5.2.6 Impaired cardiac function including any one of the following:

1. Clinically significant resting brachycardia (<50 beats per minute).
2. QTc > 450 msec on baseline ECG. If QTc >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc.
3. Myocardial infarction within 12 months prior to starting study.
4. Other clinically significant uncontrolled heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension).
5. History of or presence of clinically significant ventricular or atrial tachyarrhythmias. (including congenital long QT syndrome or a known family history of congenital long QT syndrome)

5.2.7 Allogeneic cell infusion within 100 days

5.2.8 Uncontrolled infections not responsive to antibiotics, antiviral medicines, or antifungal medicines.

5.2.9 Progressive malignant disease including post transplant lymphoproliferative disease.

5.2.10 Any secondary malignancy except basal and squamous cell carcinoma of the skin within the past five years.

5.2.11 Nilotinib intolerance or hypersensitivity. 5.2.12 Impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection or gastric bypass surgery).

5.2.13 Acute or chronic pancreatic disease 5.2.14 Major surgery within 4 weeks prior to Day 1 of the study or who have not recovered from prior surgery.

5.2.15 Subject is pregnant, breast-feeding, or of childbearing potential without a negative serum or urine pregnancy test within 7 days of enrollment. Male or female patients of childbearing potential unwilling to use effective contraceptive precautions throughout the trial.

5.2.16 Subject not willing to comply with treatment or response evaluation (including associated procedures such as skin biopsy).

5.2.17 Subject has a concurrent illness which in the opinion of the investigator may interfere with the treatment and evaluation of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2010-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events graded according to CTCAE v4.0 | 2 years

SECONDARY OUTCOMES:
Chronic GVHD response measured as change in physical exam and laboratory testing | baseline and 2 years
Chronic GVHD response measured as change in daily corticosteroid requirement | baseline and 2 years
Chronic GVHD response measured as frequency of treatment failure defined as discontinuation of study drug due to severe adverse effects or initiation of a new treatment for cGVHD | 2 years
Chronic GVHD response measured as change in cGVHD symptom burden | baseline and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David Miklos, Principal Investigator — Stanford University; George Chen, Principal Investigator — Stanford University
Locations (5):
- United States (4):
  - Stanford University School of Medicine, Stanford, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Roswell Park Cancer Institute, Buffalo, New York
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Gordon and Leslie Diamond Health Care Centre Hematology Administration, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Chen GL, Carpenter PA, Broady R, Gregory TK, Johnston LJ, Storer BE, Beumer JH, Qiu J, Cerda K, Le R, Otani JM, Liu H, Ross MA, Arai S, Flowers MED, McCarthy PL, Miklos DB. Anti-Platelet-Derived Growth Factor Receptor Alpha Chain Antibodies Predict for Response to Nilotinib in Steroid-Refractory or -Dependent Chronic Graft-Versus-Host Disease. Biol Blood Marrow Transplant. 2018 Feb;24(2):373-380. doi: 10.1016/j.bbmt.2017.10.021. Epub 2017 Oct 16. PMID 29051021